CLINICAL TRIAL: NCT06508723
Title: Long-term Clinical and Radiographic Comparison of Dental Implants with Different Surface Properties Placed in the Posterior Region
Brief Title: Comparison of Dental Implants with Different Surface Properties
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, assoc.prof.dr., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-03/04
Record Dates: First submitted 2024-07-15; First posted 2024-07-18 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Dental Implant Failed; Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: randomized, controlled, prospective
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Other): The group in which implants with a Ti-Ultra surface are placed.
  Interventions: Procedure: Dental implant placement
- Control Group (Other): The group in which implants with a Ti-Unite surface are placed.
  Interventions: Procedure: Dental implant placement

INTERVENTIONS:
Procedure: Dental implant placement — The same routine implant placement protocol will be applied to both study groups with different surfaces and will be placed in the bone. After local anesthesia, a full-thickness flap will be raised. The implant socket will be created according to the protocol recommended by the company and all implants will be placed in the socket with a torque force of 35 N and the implants will be placed. Once bleeding control is achieved, the flap will be closed primarily. Healing caps will be installed after 3 months. After waiting for wound healing, prosthetic restoration will be performed.

SUMMARY:
This controlled, parallel clinical study aims to compare the effect of fixed prosthetic restorations placed in the posterior region with different implant surfaces on clinical and peri-implant marginal bone loss.

The main question(s) it aims to answer are:

Is there a difference between peri-implant marginal bone loss levels in dental implants with two different surfaces placed in the posterior region? Is there a difference in peri-implant clinical parameters in dental implants with two different surfaces placed in the posterior region? The study includes a test group (implant with Ti-Ulta surface) and a control group (implant with Ti-Unite surface).

Two implants with different surfaces will be placed in the bone following the same routine implant placement protocol.

DETAILED DESCRIPTION:
Dental implants have become one of the most common treatments used for the rehabilitation of lost teeth. Dental implant surfaces have been roughened in different ways to increase the degree of osseointegration. A recent review reported that five different types of implant surfaces have been documented over more than 10 years. These surfaces were evaluated in 5 parts: machined, titanium plasma spray (TPS), sprayed, SLA (sandblasted and acid-etched), and anodized. The properties of an implant surface have long been identified as an essential factor in achieving and maintaining osseointegration. Modifications made to the implant body surface aim to support osseointegration and the reduction of bacterial adhesion. Pathogenic microbial colonization can lead to peri-implantitis and peri-implant marginal bone loss, resulting in dental implant failure. Roughness, porosity, and surface chemistry are essential factors for osseointegration. In particular, surface chemistry is vital in increasing cell adhesion.

An example of those produced by rearrangement of the outermost surface layer is the Ti-Unite (Nobel Biocare AG, Zurich, Switzerland) implant, where the oxide thickness is increased, and an anodizing process breaks the boundary between titanium crystals. Ti-Unite was introduced in 2001 and is among the best-selling dental implant surfaces worldwide. Nowadays, the Ti-Ultra (Nobel Biocare AG, Zurich, Switzerland) surface structure is being introduced. This redesigns the surface chemistry and topography to optimize tissue integration at all implant levels. Ti-Ultra is an ultra-hydrophilic, multizone, anodized implant surface with a graduated surface from implant neck to apex. There are studies in the literature comparing different implant surfaces.

The aim of this study is to compare the effects of fixed prosthetic restorations placed in the posterior region with different implant surfaces on clinical and peri-implant marginal bone loss.

The study will be carried out by Kütahya Health Sciences University, Faculty of Dentistry, Department of Periodontology. Systemically healthy patients between the ages of 18 and 99 and patients who have missing teeth in the posterior region and want to have a restoration with a dental implant will be included. Patients will be evaluated in two different groups: test and control groups. Patients were assigned to study groups. It will be distributed randomly and with a sealed envelope method. While dental implants with a Ti-Ultra surface will be included in the test group, dental implants with a Ti-Unite surface will be placed in the control group. All patients will undergo implant surgery and prosthetic restorations with the protocol recommended by the same company. After functional loading, patients will be followed for 12 months and routine clinical evaluations will be performed. Measurements and radiographic examinations will be obtained.

Before the operation, systemic and dental anamnesis will be taken from the patients and clinical measurements will be recorded. Periodontal indices such as plaque index, gingival index, bleeding on probing index and pocket depth will be recorded in both implant groups. Before the operation, the patient's bone amount will be evaluated on cone beam computed tomography and planning will be made. In both implant groups, keratinized mucosal thickness, keratinized mucosal height and vertical mucosal height will be measured in the area where the implant will be placed. Before and during the dental implant treatment operation, mesial, distal, buccal and lingual-palatal bone thickness measurements of the implant socket will be made with a digital caliper. Post-operative (T0), post-prosthetic loading (T1), 6th month (T2) and 1st year (T3) periapical x-rays will be taken. The amount of peri-implant marginal bone loss will be evaluated using software on standardized control periapical radiographs to be taken at the end of one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

Please find below the revised text which is clearer and free of any spelling, grammar or punctuation errors:

1. The patient must be between the ages of 18 to 99 years.
2. The patient should not have any systemic diseases.
3. There must be a toothless area in either the mandibular or maxillary region.
4. There must be natural teeth present in the opposing arch.
5. The patient should be periodontally healthy.
6. There should not be any oral or mucosal diseases present.
7. There must be sufficient bone present for implant placement, with a diameter of at least 3.5 mm and a height of 8 mm.

Exclusion Criteria:

Please find below a list of factors that may affect dental treatment and require special consideration:

1. Patients who fall outside the specified age range.
2. Patients with systemic diseases.
3. Patients who have received radiotherapy to the head and neck region.
4. Patients who have bruxism habits.
5. Patients who smoke more than 10 cigarettes per day.
6. Patients who use drugs that suppress the immune system or impair healing, such as steroids or bisphosphonates.
7. Patients with alcohol and substance addiction.
8. Patients who do not comply with treatment.
9. Pregnant women and those who are breastfeeding.
10. Mentally retarded patients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Peri-implant marginal bone loss | 1-year follow-up of all implants after prosthetic loading
  The primary outcome was the assessment of marginal bone loss on radiographs at 1-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Guler Ayyildiz, Principal Investigator — Kutahya Health Science University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If contacted, the principal researcher's evaluation will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after the study is completed and published
Access Criteria: If contacted, the principal researcher's evaluation will be shared.